CLINICAL TRIAL: NCT05900401
Title: Delayed Tolerance Through Mixed Chimerism
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ossium Health, Inc. (Industry); ITB-Med LLC (Industry)
Responsible Party: Principal Investigator, Tatsuo Kawai, MD, PhD, MD, PhD -- Professor of Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P000486
Record Dates: First submitted 2023-05-18; First posted 2023-06-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure; Kidney Transplant; Complications; Chimera
Keywords: Tolerance; Transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Bone Marrow Transplantation; fludarabine; Cyclophosphamide; Rituximab; siplizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kidney and Stem Cell Recipients (Experimental): Months-Years after standard transplant, patients will undergo bone marrow transplant (either from prospective collection of stem cells from their living donor, or from bone marrow collected at the time of deceased donation)
  Interventions: Other: Bone Marrow Transplant; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Siplizumab
- Kidney and Stem Cell Donors (Experimental): PBSC will be collected from the LD via leukapheresis 1-4 weeks before the scheduled HSCT. The donor will first undergo standard GCSF mobilization: GCSF (can be TBO-GCSF) dosed at 10 mcg/kg/d (rounded to nearest pre-filled syringe) administered subcutaneously daily for 5 consecutive days. On the 5th day, the donor will undergo standard large volume leukapheresis. The target yield will be 2-3 x 106 CD34+ cells / kg of actual recipient body weight. A maximum of 3 days of pheresis will be allowed. A minimum of 2 x 106 CD34+ cells / kg of actual recipient body weight will be required to proceed
  Interventions: Procedure: Peripheral Blood Stem Cell Collection

INTERVENTIONS:
Other: Bone Marrow Transplant — Months-Years after standard transplant, patients will undergo bone marrow transplant (either from prospective collection of stem cells from their living donor, or from bone marrow collected at the time of deceased donation)
  Arms: Kidney and Stem Cell Recipients
Procedure: Peripheral Blood Stem Cell Collection — PBSC will be collected from the LD via leukapheresis 1-4 weeks before the scheduled HSCT. The donor will first undergo standard GCSF mobilization: GCSF (can be TBO-GCSF) dosed at 10 mcg/kg/d (rounded to nearest pre-filled syringe) administered subcutaneously daily for 5 consecutive days. On the 5th day, the donor will undergo standard large volume leukapheresis. The target yield will be 2-3 x 106 CD34+ cells / kg of actual recipient body weight. A maximum of 3 days of pheresis will be allowed. A minimum of 2 x 106 CD34+ cells / kg of actual recipient body weight will be required to proceed.
  Arms: Kidney and Stem Cell Donors
Drug: Fludarabine — Fludarabine 15 mg/m2/day on days -5 to -3 (3 doses)
  Arms: Kidney and Stem Cell Recipients
Drug: Cyclophosphamide — Cyclophosphamide (CP) 30 mg/kg/day on days -5 and -4
  Arms: Kidney and Stem Cell Recipients
Drug: Rituximab — Rituximab on study day -6
  Arms: Kidney and Stem Cell Recipients
Drug: Siplizumab — Siplizumab (anti-CD2 mAb) on days, -2, -1, 0 and +1.
  Arms: Kidney and Stem Cell Recipients

SUMMARY:
This study will examine the safety and effectiveness of a bone marrow transplant after kidney transplant (from either a living or deceased donor). An investigational medication and other treatments will be given prior to and after the transplant to help protect the transplanted kidney from being attacked by the body's immune system

DETAILED DESCRIPTION:
Recipients of previous living donor (LD) or deceased donor (DD) kidney transplants that were maintained on conventional immunosuppression (I.S.), will receive a conditioning regimen that includes rituximab on study day -6, fludarabine 15 mg/m2/day on days -5 to -3 (3 doses), Cyclophosphamide (30 mg/kg/day) on days -5 and -4, followed by local thymic irradiation (7 Gy) on day -1 and Siplizumab (anti-CD2 mAb) on days, -2, -1, 0 and +1. Donor hematopoetic stem cells (HSCs) will be infused on study day 0. Methylprednisolone 250mg/day will be started on day 0 and tapered off by day 20 (Fig. 2). Prophylaxis will be provided for hemorrhagic cystitis, PCP, fungal infection, CMV, and perioperative infection. All patients who require any blood transfusion will receive only leukocyte-depleted and irradiated blood products for a period of at least 12 months following HSC Transplant. The recipients will undergo renal allograft biopsy at 6 months after HSCT. If the I.S. withdrawal criteria are met, I.S. will be slowly tapered off by 9-12 months

ELIGIBILITY:
Recipient Inclusion Criteria

1. Male or female 18-65 years of age.
2. Kidney transplant recipients from either LD or DD, with cryo-preserved HSCs available, good renal function (GFR>60 ml/min/1.73m2), normal current allograft biopsy, and no history of documented rejection episodes.
3. First or second renal transplant.
4. Use of FDA-approved methods of contraception (those with less than a 3% failure rate) by all recipients from the time that study treatment begins until 104 weeks (24 months) after renal transplantation. (For further information on FDA- approved methods of contraception, see https://www.fda.gov/media/150299/download
5. Ability to understand and provide informed consent.
6. Negative COVID-19 test during screening and two days prior to HSC transplantation (HSCT).

Deceased Donor (DD)

1. Male or female 18-70 years of age.
2. Consent to donate vertebral bones is obtained from the donor family.
3. HSCs are successfully cryopreserved and saved >2X106/kg (CD34+ cells) of the recipient.
4. Acceptable laboratory parameters (hematology in normal or near-normal range. Liver function <2 times the upper limit of normal, and normal creatinine)
5. Negative for viral infection with HbsAg, HIV, HCV, or HTLV-1
6. Negative COVID-19 test at the time of HSC procurement.

Living Donor (LD)

1. Willingness to provide HSCs by leukapheresis or bone marrow aspiration.
2. Negative serologic pregnancy test for females of childbearing potential
3. Good general health as per conventional evaluation for kidney donation.
4. Acceptable laboratory parameters (hematology in normal or near normal range. Liver function <2 times the upper limit of normal, and normal creatinine)
5. Negative for viral infection with HbsAg, HIV, HCV, or HTLV-1.
6. Cardiac/pulmonary function within normal limits (CXR, ECG).
7. Ability to understand and provide informed consent.
8. Meets standard institutional criteria for PBSC collection.
9. Negative COVID-19 test during screening and two days prior to PBSC collection.

Recipient Exclusion Criteria

1. ABO blood group-incompatible renal allograft.
2. Evidence of anti-HLA antibody (donor specific with an MFI >1000) as assessed by routine methodology (Luminex)
3. Previous history of biopsy proven rejection.
4. Persistent Leukopenia (WBC less than 2,000/mm3) or thrombocytopenia (<100,000/mm3).
5. Seropositivity for HIV-1, hepatitis B surface or core antigen, or hepatitis C virus (confirmed by hepatitis C virus RNA).
6. Active infection
7. Left ventricular ejection fraction < 40% as determined by TTE or clinical evidence of heart failure.
8. Forced expiratory volume FEV1 or DLCO < 50% of predicted.
9. Lactation or pregnancy.
10. History of cancer (following the American Transplant Society Guidelines)
11. Underlying renal disease etiology with high risk of disease recurrence in the transplanted kidney (such as focal segmental glomerulosclerosis). Autoimmune diseases such as Lupus and Thrombotic Thrombocytopenic Purpura.
12. Enrollment in other investigational drug studies within 30 days prior to enrollment.
13. Abnormal (>2 times lab normal) values for (a) liver function chemistries (ALT, AST, AP), (b) bilirubin, (c) coagulation studies (PT, PTT), or any patients on chronic anticoagulation therapy.
14. Allergy or sensitivity to any component of Siplizumab, fludarabine, CP, tacrolimus, MMF or rituximab.
15. Any medical condition that the investigator deems incompatible with participation in the trial. This includes a history of alcohol abuse or illicit drug use/dependence.
16. Non-insulin dependent diabetes (NIDDM) without good blood glucose control (HbA1c<7). Severe retinopathy, gastroparesis, or severe neuropathy which prevent subject's normal independent daily activities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of transient mixed chimerism | 3 months
Incidence of renal allograft tolerance | 2 years after immunosuppression withdrawal

SECONDARY OUTCOMES:
Incidence of Participant Survival | 2 years after immunosuppression withdrawal
Incidence of Graft Survival | 2 years after immunosuppression withdrawal
Incidence of Chimeric Transition Syndrome | 3 months
Incidence of Allograft Rejection | 2 years after immunosuppression withdrawal
  Measuring incidence of acute or chronic rejection free survival
Incidence of DSA | 2 years after immunosuppression withdrawal
Incidence of GvHD | 2 years after immunosuppression withdrawal
Incidence of infections | 2 years after immunosuppression withdrawal
  Clinically significant, invasive or resistant opportunistic infection
Incidence of thymic irradiation toxicities | 2 years after immunosuppression withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kawai, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided